CLINICAL TRIAL: NCT01622010
Title: The Effects of DVD Education on Physical Activity and Self Management of Heart Failure: A Randomized Controlled Trial
Brief Title: The Effects of DVD Education on Physical Activity and Self Management of Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There is a lower recruitment rate than projected.
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Kelly Waters, Senior Physiotherapist, St. Boniface Hospital, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2012:101
Record Dates: First submitted 2012-05-22; First posted 2012-06-18 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Patient Education as Topic; Physical Therapy Specialty
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care with video enhancement (Experimental): Receive standard care of an invitation to attend an Allied Health Education Class. May be referred to physiotherapy from Heart Failure Clinic at Physician request per standard clinic protocol. In addition are provided a copy of "Keeping the Beat with Physiotherapy: Heart Failure edition" education DVD related to heart failure, exercise and self management.
  Interventions: Behavioral: Allied Health Education Class Option; Other: Physiotherapy treatment intervention on referral; Device: Keeping the Beat with Physiotherapy: Heart Failure edition
- Standard care (Active Comparator): Receive standard care of an invitation to attend an Allied Health Education Class. May be referred to physiotherapy from Heart Failure Clinic at Physician request per standard clinic protocol.
  Interventions: Behavioral: Allied Health Education Class Option; Other: Physiotherapy treatment intervention on referral

INTERVENTIONS:
Behavioral: Allied Health Education Class Option — An Allied Health Education Class is provided as part of standard care on an optional basis. It involves a one time attendance at a 90 minute class which provides basic education from a multidisciplinary team.
Other: Physiotherapy treatment intervention on referral — The option exists for referral to physiotherapy, according to standard protocol, for assessment and individual exercise prescription.
Device: Keeping the Beat with Physiotherapy: Heart Failure edition — Educational DVD covering the basics of physiotherapy education for the patient with heart failure.
  Arms: Standard care with video enhancement

SUMMARY:
The purpose of this research is to determine if there is a greater behaviour change in self management of heart failure following reinforced multimedia education focusing on physical activity as compared to standard care. It is the investigators belief that participants who receive DVD education in addition to usual care will show improved self management in comparison to receiving usual care alone. The investigators anticipate fewer hospital admissions due to improved self care management.

DETAILED DESCRIPTION:
With an aging population, heart failure is becoming more common and there is an increasing role for physiotherapy involvement with these patients. The Heart Failure Clinic is conducted by a heart failure physician, cardiac nurse, and a pharmacist. Occupational and Physical Therapists are available on a consult basis. The Clinic has expanded quickly from 49 new patients in 2004 - 2005 to 435 new patients in 2010 - 2011.

Due to space and time constraints in the clinic an Allied Heath Education Class was created to provide an interactive multidisciplinary education session. All new patients, regardless of their NYHA classification, and their families are invited to attend the class. Speakers include a Physiotherapist, Occupational Therapist, Dietician and Pharmacist. There is a didactic section followed by discussion after each of the speakers.

Few studies have focused on physical activity as one of the major self management strategies for heart failure. There is little understanding by patients about how physical activity can improve symptoms of heart failure over time in conjunction with other lifestyle modifications. Physiotherapists have the skills to provide this education and develop individual exercise programs. Patients are currently provided with verbal and written educational material regarding a diagnosis of heart failure, physical activity, diet and medication.

Previous experience with patients following acute cardiac events, either medical or surgical, has shown that providing patients with a DVD which reinforced inpatient education was successful in bridging the gap between inpatient and outpatient rehabilitation programs. Patients were able to review the education provided in their own time. Therefore, a DVD was developed which focused on typical education provided to the heart failure patient by the physiotherapist.

We will compare two randomly assigned groups. The first will receive standard education received in heart failure clinic and an optional Allied Health Education Class plus a copy of the Keeping the Beat with Physiotherapy: Heart Failure edition DVD. The second group will receive the standard education provided through the heart failure clinic and the optional education class.

Participants will be followed up three times over a six month period via telephone. The survey questions require a simple yes/no answer or are of a likert-style. After each telephone survey participants, will be asked to mail in their exercise and weight logs. Chart reviews will also be conducted for the collection of readmission rates and the number of clinical visits occurring during the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart failure
* Attending Heart Failure Clinic for the first time
* New York Heart Association Classification - any

Exclusion Criteria:

* Inability to understand English or French well enough to participate in a telephone survey
* Being worked up for transplant, ventricular assist device or other form of cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Waters, BMR (PT), Principal Investigator — St. Boniface Hospital; Heather J Christie, BMR(PT), MSc, Study Chair — St. Boniface Hospital; Jenn Rybuck, BMR(PT), Study Chair — St. Boniface Hospital
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care With Video Enhancement | Standard Care
Started | 18 | 12
Completed | 12 | 8
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care With Video Enhancement | Standard Care | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (16.2) | 65.7 (7.0) | 63.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 15 | 12 | 27
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 12 | 30
New York Heart Association (NYHA) Classification [Number; unit: participants] — NYHA Classification:
  Class I: No limitation of physical activity Class II: Slight limitation of physical activity, ordinary physical activity leads to fatigue, palpitation, dyspnea, or anginal pain; comfortable at rest Class III: Marked limitation of physical activity, less-than-ordinary activity results in fatigue, palpitation, dyspnea, or anginal pain; comfortable at rest Class IV: Inability to carry on any physical activity without discomfort but also symptoms of heart failure or the anginal syndrome even at rest, with increased discomfort if any physical activity is undertaken
  participants
    NYHA class I | 4 | 4 | 8
    NYHA class II | 4 | 4 | 8
    NYHA class III | 9 | 3 | 12
    NYHA class IV | 0 | 0 | 0
    Unclassified | 1 | 1 | 2
Working Status [Number; unit: participants]
  Retired | 6 | 3 | 9
  Disability | 1 | 0 | 1
  Working | 5 | 2 | 7
  Unknown | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Exercise - General
Description: Based on telephone survey responses - ranked Likert scale, 1 - 4 with 1 representing the better outcome
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Standard Care With Video Enhancement | Standard Care
Number analyzed (Participants) | 17 | 9
participants
  Daily | 6 | 3
  Few times a week | 5 | 5
  Few times a month | 1 | 0
  Not at all | 5 | 1
Statistical Analysis 1: Comparison: Standard Care With Video Enhancement vs Standard Care; Test type: Equivalence — P value 0.05 used; p = 0.487, Chi-squared

2. Secondary Outcome: Readmission Rate
Description: Collected from telephone survey and chart review
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Standard Care With Video Enhancement | Standard Care
Number analyzed (Participants) | 17 | 9
participants | 7 | 4

3. Secondary Outcome: Confidence in Activity Related Decision Making
Description: Based on telephone survey responses - ranked Likert scale - 1 - 4 with 1 representing better outcome
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Standard Care With Video Enhancement | Standard Care
Number analyzed (Participants) | 17 | 9
participants
  Very Confident | 4 | 2
  Confident | 10 | 4
  Somewhat confident | 2 | 2
  Not at all confident | 1 | 1
Statistical Analysis 1: Comparison: Standard Care With Video Enhancement vs Standard Care; Null hypothesis: Standard care is better than standard care with video enhancement; Test type: Non-Inferiority or Equivalence — a non-inferiority margin calculation was not performed for this study prior to its start; p = 0.628, Fisher Exact

4. Secondary Outcome: Confidence in Decision Making Regarding Weight Changes
Description: Based on telephone survey responses - with option of "Yes", "No", "Unsure" where Yes is indicative of a better outcome.
Time Frame: 3 months
Population: Do you know what to do if weight is changing?
Measure: Number; unit: participants
Groups:
- Standard Care With Video Enhancement: Allied Health Education Class Option
  Physiotherapy treatment intervention on referral
  Keeping the Beat with Physiotherapy: Heart Failure edition: Educational DVD
- Standard Care: Allied Health Education Class Option
  Physiotherapy treatment intervention on referral
Arm/Group | Standard Care With Video Enhancement | Standard Care
Number analyzed (Participants) | 17 | 9
participants
  Yes | 11 | 5
  No | 3 | 1
  Unsure | 3 | 3
Statistical Analysis 1: Comparison: Standard Care With Video Enhancement vs Standard Care; Test type: Equivalence — P Value 0.05 used; p = 0.647, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months following recruitment
Arm/Group | Standard Care With Video Enhancement | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12
Other Adverse Events (participants affected / at risk) | 0/18 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No